CLINICAL TRIAL: NCT01121315
Title: A Retrospective Epidemiological Study to Investigate Outcome and Mortality With Glucose Lowering Drug Treatment in Primary Care
Brief Title: A Retrospective Study of Cardiovascular Events Related to the Use of Glucose Lowering Drug Treatment in Primary Care
Acronym: ROSE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CSE-DUM-2010/1
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Type II
Keywords: Epidemiological; Diabetes; Glucose Lowering Drug Treatment in Primary care; CVD
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Diabetes type II patients, according to medical records, prescriptions or lab results, followed for >6 months after diagnosis.

SUMMARY:
To describe the type II diabetes population in primary care with special reference to treatment, other diseases and mortality during the last decade. To test the hypothesis that the type or combination of per oral glucose lowering drugs have different effects on the risk of cardiovascular disease and diabetic complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type II diabetes, according to medical records, diagnosis, prescription or lab assessments

Exclusion Criteria:

* Patients followed by physician for less than 6 months after diagnosis of Diabetes type II

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible subjects are all type II diabetes patients, found in medical records at the participating centres. Patient data from the period 1 January 1999 - 31 December 2009 will be included in the observation. To ensure a representative selection of primary care centers, selection of study sites will be based on the following criteria to ensure a representative sample of the Swedish population: a mix of rural and urban areas, public and private care providers, small, mid sized and large primary care centers.
Sampling Method: Non-Probability Sample
Enrollment: 58326 (Actual)
Dates: Start 2010-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Composite end-point consisting of Cardiovascular Disease, elective coronary revascularisation and mortality | The endpoints will be extracted from the medical records on one occassion, covering a period of one decade.

SECONDARY OUTCOMES:
Retinopathy, renal failure, hypoglycaemic episodes, other diabetic complications | The endpoints will be extracted from the medical records on one occasion, covering a period of one decade.
Time from: Metformin (MET) to Insulin (INS) versus Metformin (MET) -> Metformin (MET)+Sulfonylurea (SU) ->Insulin (INS) | The endpoints will be extracted from the medical records on one occasion, covering a period of one decade.
Number of consultations in primary care. Number of hospitalisations | The endpoints will be extracted from the medical records on one occasion, covering a period of one decade.

CONTACTS AND LOCATIONS:
Overall Officials: Leif Lohm, MD, Study Director — AstraZeneca Nordic, Södertälje; Gunnar Johansson, MD, Principal Investigator — Uppsala University, Sweden; Carl Johan Östgren, MD, Study Chair — Ödeshögs VC; Johan Sundström, MD PhD, Study Chair — Uppsala University Hospital
Locations (1):
- Research Site, Uppsala, Sweden

REFERENCES:
- [Derived] Grundvold I, Bodegard J, Nilsson PM, Svennblad B, Johansson G, Ostgren CJ, Sundstrom J. Body weight and risk of atrial fibrillation in 7,169 patients with newly diagnosed type 2 diabetes; an observational study. Cardiovasc Diabetol. 2015 Jan 15;14:5. doi: 10.1186/s12933-014-0170-3. PMID 25589001
- [Derived] Sundstrom J, Sheikhi R, Ostgren CJ, Svennblad B, Bodegard J, Nilsson PM, Johansson G. Blood pressure levels and risk of cardiovascular events and mortality in type-2 diabetes: cohort study of 34 009 primary care patients. J Hypertens. 2013 Aug;31(8):1603-10. doi: 10.1097/HJH.0b013e32836123aa. PMID 23625112
- [Derived] Ostgren CJ, Sundstrom J, Svennblad B, Lohm L, Nilsson PM, Johansson G. Associations of HbA1c and educational level with risk of cardiovascular events in 32,871 drug-treated patients with Type 2 diabetes: a cohort study in primary care. Diabet Med. 2013 May;30(5):e170-7. doi: 10.1111/dme.12145. Epub 2013 Mar 13. PMID 23350893